CLINICAL TRIAL: NCT04911439
Title: Influencia de Los Niveles de Alerta en el Aprendizaje Motor de Una Tarea Manual Precisa, en la Memoria a Corto y Largo Plazo y en la Capacidad de Imaginación Motora
Brief Title: Influence of Arousal on Motor Learning, Memory and Motor Imagery Ability in Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susana Nunez Nagy (Other)
Collaborators: University of Alcala (Other); Universidad Complutense de Madrid (Other); European University of Madrid (Other); Claude Bernard University (Other)
Responsible Party: Sponsor-Investigator, Susana Nunez Nagy, PhD. Associate Professor of Physiotherapy, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEID/HU/2021/1/011
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Arousal
Keywords: Arousal; Motor Learning; Memory; Motor Imagery Ability

STUDY DESIGN:
Intervention Model Description: As participants complete the State-Trait Anxiety Inventory, and are found to be free of trait anxiety, and state anxiety, they will be randomised in parallel to one of the three intervention groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant does not know what the other participants are doing, the researcher knows which study and group the subject is in, but only sets up the computerized presentations for each group and assigns folders within the computer that collects the data, thus avoiding a possible information bias, and finally, another researcher blind to the intervention will analyse the data to obtain the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Arousal (Active Comparator): This group will see 25 affective images of the International Affective Picture System with low arousal level during 8-12 randomly seconds each one at time and with randomly rest of 8-12 seconds between images.
  Interventions: Other: Low Arousal
- Medium Arousal (Active Comparator): This group will see 25 affective images of the International Affective Picture System with medium arousal level during 8-12 randomly seconds each one at time and with randomly rest of 8-12 seconds between images.
  Interventions: Other: Medium arousal
- High Arousal (Active Comparator): This group will see 25 affective images of the International Affective Picture System with high arousal level during 8-12 randomly seconds each one at time and with randomly rest of 8-12 seconds between images.
  Interventions: Other: High arousal

INTERVENTIONS:
Other: Low Arousal — This group will see affective images of the International Affective Picture System with low arousal level
  Arms: Low Arousal
Other: Medium arousal — This group will see affective images of the International Affective Picture System with medium arousal level
  Arms: Medium Arousal
Other: High arousal — This group will see affective images of the International Affective Picture System with high arousal level
  Arms: High Arousal

SUMMARY:
In motor learning is essential to consider that movements are produced by the cooperation and combination of many brain structures and are influenced by the emotions to which individuals are subjected. Several neural circuits have been identified that closely link the emotional system and the motion control system.

Arousal is associated with many emotional responses and has effects on the nervous and motor system. In line with the "Inverted 'U' Hypothesis", all levels of both high and low arousal do not allow optimal task performance, yet moderate levels lead to excellent performance. Arousal also plays a vital role in movement learning, where a critical element is memory. There is evidence that a minimum level of arousal is required to encode or record information and that that moderate levels of arousal improve memory.

Understanding how movement, emotions and interactions are regulated is significant because of the large number of movements humans perform. Of these, manual tasks represent precise movements that require the integration of many elements by the nervous system to perform these tasks successfully. How different levels of arousal influence the way manual tasks are learned is still unknown.

On the other hand, motor imagery (MI) is a cognitive process that is an important contributor to how movements are planned and executed. The use of MI has been recommended to improve movement learning and task execution. For an effective and individualize MI program is imperative to know this capacity. However, how different levels of arousal can affect our motor imagery ability is also still unknown.

The main objective of this study is to determine and quantify the effects of arousal levels in the learning of a precise manual task not previously trained on four parameters of fine motor control: time, error, speed, and accuracy. On the other hand, the aim is to determine if the ability of internal visual, external visual, and kinaesthetic imagery varies when participants are subjected to different levels of arousal.

Researches expect that non-anxious, non-stressed participants who are shown images that elicit an optimal level of arousal will show better motor performance on the fine motor task and better motor imagery ability. In contrast, researches expect that participants without anxiety and stress who are shown pictures that elicit a sub-optimal level of arousal will show poorer motor performance on the fine motor task and poorer motor imagery ability.

DETAILED DESCRIPTION:
In order to meet the study objectives of determining and quantifying the effects of arousal levels on learning a precise manual task and on motor imagery ability, this study will be conducted. The development of the study will take place in a conditioned room belonging to the University of Alcala, the Complutense University of Madrid, or the European University of Madrid. The study may also be carried out in other Spanish and international university centers, subject to the consent and permission of the respective centres. The study will be carried out by all national and international laws, regulations, and recommendations.

The study design will be longitudinal, experimental, randomized, and double-blind, as specified in the present registry.

The study population will be composed of participants who are undergraduate and postgraduate students at the university centers where the study will be carried out, from which the participants will be recruited. All participants included in the study must meet the study selection criteria and participate voluntarily after reading the information sheet and signing the informed consent form.

The study will consist of three intervention groups, in which low, medium, or high arousal will be induced, respectively. Each group will consist of a minimum number of 30 subjects to be able to study the desired effect.

After each participant freely chooses to participate in the study, an initial questionnaire will be administered to ensure that each participant meet the criteria for inclusion in the study. At this point, the participant will be coded and assigned a number, which will serve as identification throughout the study. Participants will take the State-Trait Anxiety Inventory (STAI), one of the most widely used instruments for the self-reported assessment of anxiety and equivalent to a measure of stress, as it considers the amount of stressful stimulus. Thus, the two components of anxiety will be assessed: state anxiety and trait anxiety. Participants with scores indicative of state or trait anxiety will be excluded from the study, and those with scores indicating neither trait anxiety nor state anxiety will be included. Included participants will be randomized through sealed envelopes stratified by gender to one of three experimental groups: low arousal, medium arousal, and high arousal. Participants will also take the Movement Imagery Questionnaire-3 (MIQ-3) to measure internal visual, external visual, kinaesthetic imagery ability, and the Edinburgh Handedness Inventory (EHI) to determine the participant's laterality. Depending on the group to which participants have been assigned, participants will be visualize a series of International Affective Picture System (IAPS) images that will induce the different states of arousal. The IAPS is one of the most widely used standardized emotion-eliciting stimulus sets in experimental research and has been shown to produce reliable and measurable changes in all three emotional response systems in the study population of this study: subjective-verbal, behavioral and physiological. After visualizing the images, participants will learn a precise manual task with the non-dominant hand. The task will consist of going over a 127 mm circumference on a graphics tablet at a rate of 2 seconds per lap, which will be set by a metronome using a wireless pen that will leave no trace of ink but will store the data in the MATLAB program via the graphics tablet. Thus, data from the learning process and short-term memory of the task will be recorded. Afterward, there will be a 20-minute break during which participants will perform the MIQ-3 again. Finally, the task data will be collected to record the long-term memory of the manual task.

In addition, during all experiments, electrodermal activity and heart rate variability will be recorded using the Empatica E4 physiological variable measurement wristband. This measurement of physiological variables will serve to confirm that a significant emotional effect has been generated and to test motor imagery processes since both arousal and motor imagery produce activation of the autonomic nervous system.

The analysis and processing of data from MATLAB version R2020b, and the Empatica E4 wristband will be performed using SPSS 25.0 statistical software and Kubios HRV software (for HRV analysis).

First, appropriate statistical analyses will be performed to see if the data are distributed according to a standard curve through the Shapiro-Wilk test and to assess the influence of sex and age.

Subsequently, the descriptive analysis of the relative and absolute frequencies for the qualitative variables of gender and age will be carried out, and their homogeneity will be tested using the Chi-square test. The descriptive analysis of the quantitative variables of time, error, speed, accuracy, electrodermal activity, heart rate variability, and kinaesthetic, internal visual, and external visual imagery will also be carried out. If the variable conforms to the normal, the mean, range, and standard deviation shall be calculated. If the variables do not conform to normality, non-parametric tests will be performed.

Comparative analysis will be performed using mixed ANOVA to see the differences in the mean values respective to motor control (time, error, speed, and accuracy), and the differences between the first and last lap and between consecutive laps of the task in the same four parameters, both in the task performed in the short term and the long term. A further ANOVA analysis will take place for imagery ability, comparing the results obtained at the two respective points during the experiment.

The effect of learning between laps will be analyzed by repeated-measures ANOVA comparing each motor control measurement parameter with respect to the lapping factor. Electrodermal activity, and heart rate variability during the measurement of imagery ability, emotional state induction, manual task learning, and its maintenance in the short and long term will also be studied by repeated-measures ANOVA.

For hypothesis testing, a significance level of 0.05 will be set.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 35 years of age.
* Normal or corrected vision specifying the method of correction.
* Normal or corrected hearing specifying method of correction.
* Unfamiliar with the assessment and uses of motor imagery.

Exclusion Criteria:

* Subjects who have suffered fractures, dislocations, or traumatic processes in any segment of the non-dominant upper limb or fingers, wrist, or elbow of the dominant upper limb in the last 6 months.
* Subjects with learning disabilities or problems in reading or writing.
* Subjects with a history of any neurological disease, cardiovascular disease, myopathic disease, epileptic seizure, absence seizure, sleep apnoea, chronic fatigue syndrome, or fibromyalgia.
* Taking any medication to suppress anxiety, to sleep, antidepressants, antihistamines, muscle relaxants, psychotropic, or other medications that interfere with the nervous system.
* Intake of nervous system depressants or stimulants such as caffeine or theine in the last 8 hours.
* Presence of State-Trait Anxiety Inventory scores corresponding to trait anxiety and state anxiety.
* Presence of localised skin lesion or disease in the wrist area.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Manual task execution time measured in seconds by MATLAB. | During procedure
  This is the time taken by the subject to execute a complete circumference. It shall be expressed in seconds (s). It shall be recorded and measured through MATLAB.
Manual task execution error measured in seconds by MATLAB. | During procedure
  It shall be the inaccuracy committed by the subject in the tracing of the reference circumference. The dots per inch (dpi) or pixels per inch (pix) recorded in each lap from lap No. 1 to lap No. 20 shall be considered. It shall be recorded and measured by MATLAB.
Execution Speed | During procedure
  This shall be the pixels drawn per unit of time. It shall be expressed in pixels per second (pix/s). It shall be recorded and measured by MATLAB.
Execution Accuracy | During procedure
  This refers to the dispersion of the set of values obtained from repeated measurements under the same conditions of the values of each of the laps. It shall be calculated as the ratio between the number of errors made divided by the execution speed from the previous data recorded in MATLAB. It shall be expressed in seconds: No. errors (pix) /V (pix/s) = (s).
Motor Imagery Ability | Two points: Before procedure, resting period during procedure
  This will be measured using the Movement Imagery Questionnaire-3, differentiating between the kinaesthetic, external visual and internal visual imagination subscales. Each subscale has 4 items and each item can be scored on a Likert scale from 1 to 7 points, where 1=very difficult to see/feel the movement and 7=very easy to see/feel the movement. Therefore, higher scores represent greater imaginative ability and each subscale can have a minimum of 4 points and a maximum of 28 points.

SECONDARY OUTCOMES:
Latency of the Electrodermal Activity | During procedure
  The skin conductance level and skin conductance responses shall be analyzed in terms of latency (s). It shall be recorded and measured by Empatica E4 wristband.
Rise time of the Electrodermal Activity | During procedure
  The skin conductance level and skin conductance responses shall be analyzed in terms of rise time (s). It shall be recorded and measured by Empatica E4 wristband.
Amplitude of the Electrodermal Activity | During procedure
  The skin conductance level and skin conductance responses shall be analyzed in terms of amplitude (μs). It shall be recorded and measured by Empatica E4 wristband.
Heart Rate | During procedure
  The Heart Rate (Hz) shall be analyzed. It shall be recorded and measured by Empatica E4 wristband through the analysis of the Blood Volume Pulse.
Interbeat Intervals | During procedure
  The Interbeat Intervals (s) shall be analyzed. These Interbeat Intervals (IBIs) sequences will be provided by Empatica E4 wristband through the processing of the photoplethysmography signal.
Heart Rate Variability | During procedure
  The Heart Rate Variability (Hz) shall be analyzed. This measurement will be calculated from the Interbeat Intervals measured by Empatica E4 wristband through the Kubios software.

CONTACTS AND LOCATIONS:
Overall Officials: Sara T Trapero Asenjo, Master, Principal Investigator — University of Alcala; Susana N Núñez Nagy, PhD, Study Director — University of Alcala; Sara F Fernández Guinea, PhD, Study Director — Universidad Complutense de Madrid
Locations (4):
- Claude Bernard University Lyon 1, Villeurbanne, Auvergne-Rhône-Alpes, France
- Spain (3):
  - University of Alcala, Alcalá de Henares, Madrid
  - Complutense University of Madrid, Pozuelo de Alarcón, Madrid
  - European University of Madrid, Villaviciosa de Odón, Madrid

REFERENCES:
- [Background] Stins JF, Beek PJ. Effects of affective picture viewing on postural control. BMC Neurosci. 2007 Oct 4;8:83. doi: 10.1186/1471-2202-8-83. PMID 17916245
- [Background] Coombes SA, Cauraugh JH, Janelle CM. Emotion and movement: activation of defensive circuitry alters the magnitude of a sustained muscle contraction. Neurosci Lett. 2006 Apr 3;396(3):192-6. doi: 10.1016/j.neulet.2005.11.048. Epub 2005 Dec 20. PMID 16376016
- [Background] MacIntyre TE, Madan CR, Moran AP, Collet C, Guillot A. Motor imagery, performance and motor rehabilitation. Prog Brain Res. 2018;240:141-159. doi: 10.1016/bs.pbr.2018.09.010. Epub 2018 Oct 24. PMID 30390828
- [Background] Schuster C, Hilfiker R, Amft O, Scheidhauer A, Andrews B, Butler J, Kischka U, Ettlin T. Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines. BMC Med. 2011 Jun 17;9:75. doi: 10.1186/1741-7015-9-75. PMID 21682867
- [Background] Trapero-Asenjo S, Gallego-Izquierdo T, Pecos-Martin D, Nunez-Nagy S. Translation, cultural adaptation, and validation of the Spanish version of the Movement Imagery Questionnaire-3 (MIQ-3). Musculoskelet Sci Pract. 2021 Feb;51:102313. doi: 10.1016/j.msksp.2020.102313. Epub 2020 Dec 9. PMID 33310512
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Bali A, Jaggi AS. Clinical experimental stress studies: methods and assessment. Rev Neurosci. 2015;26(5):555-79. doi: 10.1515/revneuro-2015-0004. PMID 26020552